CLINICAL TRIAL: NCT00118976
Title: Optimal Dose of ACE Inhibitor for Treatment of Diabetic Nephropathy in Type 1 Diabetic Patients With Hypertension and Diabetic Nephropathy
Brief Title: Maximal Dose of Angiotensin Converting Enzyme (ACE) Inhibitor for Treatment of Diabetic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: mace
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2006-11-23 (Estimated); Status verified 2006-11

CONDITIONS: Diabetes Mellitus, Type I; Diabetic Nephropathy
Keywords: diabetic nephropathy; type 1 diabetes; albuminuria; hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies; Albuminuria; Hypertension | interventions — Lisinopril

INTERVENTIONS:
Drug: Lisinopril

SUMMARY:
The primary aim is to evaluate the anti proteinuric effect of increasing doses of the ACE inhibitor, lisinopril: 20, 40 and 60 mg daily in type 1 diabetic patients with hypertension and diabetic nephropathy.

The secondary aim is to evaluate the effect on blood pressure (24 hour ambulatory blood pressure) and kidney function (glomerular filtration rate (GFR)).

The tertiary aim is to evaluate differences in response to treatment according to ACE/insertion/deletion (ID)-genotypes and other genetic variants in the genes of the renin angiotensin system.

DETAILED DESCRIPTION:
This is a randomized, double-blind cross-over study with three treatment periods consisting of 20, 40 and 60 mg lisinopril daily in random order. The endpoints of the study will be examined after each treatment period. There is no wash out between treatment periods. To minimize the risk of hypotension every treatment period starts with 20 mg lisinopril for two weeks. Thus, the risk of adverse effects is minimized and an increase in dose from 0 mg to 60 mg lisinopril is avoided.

The patients usual antihypertensive treatments will be stopped in a period of 8 weeks (wash out) before randomization. Since diuretic drugs will be needed by almost every patient in the study to avoid oedema all patients will be treated with lasix retard 60 - 120 mg daily.

Patients:

60 type 1 diabetic patients with diabetic nephropathy and hypertension (blood pressure > 135 mm Hg systolic and/or 85 mm Hg diastolic).

Methods:

The endpoints of the study will be examined at baseline and after each treatment period corresponding to 8, 16, and 24 weeks after randomization. The following parameters are determined after each treatment period: Albuminuria (determined from three consecutive 24 hours urine collections), kidney function (GFR - by plasma clearance of 51Cr-EDTA ), and 24 hour ambulatory blood pressure (TM-2420/2421). Furthermore, the concentrations of TGF-ß, sodium, creatinine, and carbamide in the 24 hour urinary samples are determined. The plasma concentration of albumin, renin, angiotensin II, and aldosterone is measured.

DNA is extracted from a blood sample and genetic variants in the renin-angiotensin system are measured including the ACE/ID genotype.

Endpoints:

Primary endpoint: albuminuria ; Secondary endpoints: blood pressure (24 hour ambulatory) and GFR; Tertiary: differences in response to treatment in patients with different ACE/ID and other renin angiotensin system genotypes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes (WHO criteria)
* Diabetic nephropathy (2 out of 3 consecutive 24 hour urinary samples with albumin excretion > 300 mg/24hour and diabetic retinopathy in the absence of signs of other kidney or urinary tract disease) 27 or diabetic glomerulosclerosis verified by biopsy.
* Hypertension: Blood pressure > 135 mmHg systolic and/or 85 mm Hg diastolic repeatedly.
* Age from 18 to 70 years.

Exclusion Criteria:

* Age < 18 years or > 70 years.
* Pregnancy or fertile women not using adequate anticonceptive (intrauterine device, sterilization, or oral anticonceptive)
* Malignant hypertension.
* Blood pressure > 180/105 mm Hg
* Known renal artery stenosis
* GFR < 30 ml/min/1.73 m²
* Serum potassium > 4.8 mmol/ l
* Heart failure, myocardial infarction, unstable angina or coronary bypass operation within the previous three months.
* Abuse of drugs or alcohol.
* Not able to understand the written information.
* Known intolerance to ACE inhibitors.
* Chronic use of non steroid inflammatory drugs or aspirin (above 1 g/day)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-03; Study Completion 2006-09

PRIMARY OUTCOMES:
albuminuria

SECONDARY OUTCOMES:
blood pressure (24 hour ambulatory) and GFR.
Tertiary: differences in response to treatment in patients with different ACE/ID and other renin angiotensin system genotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Henrik Parving, MD, Study Chair — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Schjoedt KJ, Astrup AS, Persson F, Frandsen E, Boomsma F, Rossing K, Tarnow L, Rossing P, Parving HH. Optimal dose of lisinopril for renoprotection in type 1 diabetic patients with diabetic nephropathy: a randomised crossover trial. Diabetologia. 2009 Jan;52(1):46-9. doi: 10.1007/s00125-008-1184-8. Epub 2008 Oct 31. PMID 18974967